CLINICAL TRIAL: NCT02850978
Title: Post-marketing Surveillance (PMS) on Long-term Use of Tiotropium+Olodaterol Fixed Dose Combination (Tio+Olo FDC) 5µg/5µg in Patients With Chronic Obstructive Pulmonary Disease (Chronic Bronchitis, Emphysema) in Japan
Brief Title: Long-term Use of Spiolto Respimat in Japanese Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237.34
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Results first posted 2019-12-06 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tiotropium-olodaterol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Spiolto: Patient with COPD to received Spiolto
  Interventions: Drug: Spiolto

INTERVENTIONS:
Drug: Spiolto

SUMMARY:
Study to assess the long-term safety and effectiveness of Spiolto in Japanese patients with Chronic Obstructive Pulmonary Disease (COPD) in real-world setting

ELIGIBILITY:
Inclusion criteria:

* Patients who have been diagnosed with chronic obstructive pulmonary disease (chronic bronchitis, emphysema) by physician and need relief of various symptoms associated with Long Acting Beta2 Agonist (LABA) or Long Acting Muscarinic Antagonist (LAMA).
* Patients who are prescribed Tio+Olo FDC 5µg/5µg for the first time

Exclusion criteria:

* Patients who have been registered once in this study (i.e., re-entry of patients is not allowed).
* Patients who are participating in a registry or clinical trial.
* Patients who have a contraindication to Tio+Olo FDC 5µg/5µg defined in the package insert for Tio+Olo FDC 5µg/5µg.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1000
Sampling Method: Non-Probability Sample
Enrollment: 1335 (Actual)
Dates: Start 2016-08-23 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Multiple Locations, Japan

REFERENCES:
- [Derived] Sato A, Miyazaki A, Nakamura S. Effectiveness of Tiotropium/Olodaterol in the Real World: A Post Hoc Subgroup Analysis After the First Year of Use. Adv Ther. 2022 Oct;39(10):4692-4706. doi: 10.1007/s12325-022-02268-1. Epub 2022 Aug 10. PMID 35948844

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an observational study based on newly collected data under real-world practice in participants diagnosed with chronic obstructive pulmonary disease (COPD) (chronic bronchitis, emphysema) in Japan.
Pre-assignment Details: This non-randomized, post marketing surveillance (PMS) was a prospective study using a continuous investigation system. No specific criteria (e.g. demographic, baseline, concomitant drug in use) were defined for participant enrollment. Participants were enrolled from August 2016 to August 2017.
Groups:
- Spiolto®: Participants suffering from COPD were treated with a Fixed Dose Combination (FDC) of Tiotropium (Tio) 5 microgram (μg)/ + Olodaterol (Olo) 5 μg; solution for oral inhalation via Respimat® inhaler once daily, for 52 weeks or until discontinuation of administration.
Period: Overall Study
Arm/Group | Spiolto®
Started (Strated are registered) | 1335
Case Report Form (CRF) Collected | 1308
Treated | 1308
Completed | 909
Not Completed | 426
Not completed — Uncollectable CRF | 27
Not completed — No visit since the first visit | 35
Not completed — Adverse Event | 81
Not completed — Lack of Efficacy | 40
Not completed — Improvement in condition | 34
Not completed — Lost to Follow-up | 121
Not completed — Reason not listed | 88

BASELINE CHARACTERISTICS:
Population: Safety set: This patient set includes all patients who were documented to have taken at least one dose of Spiolto® Respimat® excluding no visit after Spiolto® Respimat® administration.
Arm/Group | Spiolto®
Number analyzed (Participants) | 1273
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206
  Male | 1067
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Drug Reactions
Description: Percentage of participants with adverse drug reactions (ADR). An adverse drug reaction (ADR) is defined as an adverse event (AE) for which either the investigator or the sponsor (or both) assess the causal relationship to Spiolto® Respimat® as "Yes".
Time Frame: From the first drug administration until 21 days after the last drug administration, up to approximately 82 weeks.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants (%)
Arm/Group | Spiolto®
Number analyzed (Participants) | 1273
Percentage of participants (%) | 3.93

2. Secondary Outcome: Change of COPD Assessment Test (CAT) Score From Baseline to Week 12
Description: The COPD Assessment Test™ (CAT) is a short 8-item questionnaire for assessment and monitoring of COPD health status in routine practice. Its scale is 0-40 (high score = poor health). The CAT questionnaire has the advantage of a reduced number of items and could be used to assess the effects of inhaled therapies. The CAT score was the sum of the values corresponding to the answers to the eight questions.
Time Frame: Baseline and Week 12
Population: Effectiveness set: The effectiveness set included all patients in the safety set except for those patients who had no any values of CAT, Forced Expiratory Volume in one second (FEV1) and Forced Vital Capacity (FVC) after Spiolto® Respimat® administration.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Spiolto®
Number analyzed (Participants) | 1255
Unit on a scale | -3.7 (7.1)

ADVERSE EVENTS:
Time Frame: From the first drug administration until 21 days after the last drug administration, up to approximately 82 weeks.
Arm/Group | Spiolto®
All-Cause Mortality (participants affected / at risk) | 38/1273
Serious Adverse Events (participants affected / at risk) | 94/1273
Other Adverse Events (participants affected / at risk) | 0/1273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spiolto® (N=1273)
Anaemia (Blood and lymphatic system disorders) | 2
Cardiac failure (Cardiac disorders) | 5
Cardiac failure congestive (Cardiac disorders) | 3
Cardio-respiratory arrest (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrioventricular block second degree (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure chronic (Cardiac disorders) | 1
Cardiovascular disorder (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Right ventricular failure (Cardiac disorders) | 1
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1
Adrenocortical insufficiency acute (Endocrine disorders) | 1
Thyrotoxic crisis (Endocrine disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Death (General disorders) | 4
Sudden death (General disorders) | 2
Pyrexia (General disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 12
Respiratory tract infection (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Infectious pleural effusion (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 3
Femur fracture (Injury, poisoning and procedural complications) | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1
Compression fracture (Injury, poisoning and procedural complications) | 1
Shunt occlusion (Injury, poisoning and procedural complications) | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1
C-reactive protein increased (Investigations) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral infarction (Nervous system disorders) | 2
Dementia (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 12
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 7
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Aortic dissection (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The study was conducted in an unblinded manner and without controls. The explanatory power of the study results was limited and the study results should be interpreted with the necessary caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/78/NCT02850978/SAP_000.pdf
  • Study Protocol (2016-05-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT02850978/Prot_001.pdf